CLINICAL TRIAL: NCT02435576
Title: Standard Follow-up Program (SFP) for Head and Neck Cancer Patients Treated With Curative Primary or Postoperative Radiotherapy or Chemoradiation (SFP Head & Neck)
Brief Title: Standard Follow-up Program (SFP) for Head and Neck Cancer Patients
Acronym: H&NTOX
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SFP2007-03
Record Dates: First submitted 2015-03-27; First posted 2015-05-06 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Cancer
Keywords: Acute toxicity; Late toxicity; NTCP models; Proton therapy; Patient-rated outcomes; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy; Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiotherapy (primary or postoperative)

SUMMARY:
The primary and general objective of the clinical introduction of the SFP as the current standard of care is to improve the quality of radiotherapy for head and neck cancer patients by reducing radiation-induced side effects without hampering treatment efficacy in terms of locoregional tumour control and overall survival and to systematically evaluate the beneficial effect of newly introduced radiation technology for this particular group of patients. The clinical introduction of the SFP will allow for a systematic and broad scale quality improvement cycle for head and neck cancer patients treated with radiotherapy. In fact, this methodology can be considered a kind of quality circle for the clinical introduction of new radiation techniques, aiming at continuous efforts for further improvement.

DETAILED DESCRIPTION:
Specific objectives

* To develop, validate, and improve normal tissue complication probability (NTCP) models for a wide variety of acute and late radiation-induced side effects relevant for head and neck cancer patients (step 1);
* To use the outcome of the NTCP models to better inform patients on the risks on acute and late toxicity;
* To use the outcome of the NTCP models for the definition of dose constraints for radiotherapy treatment planning in current practice;
* To use the outcome of the NTCP models for the development and investigation of the potential benefit of new and emerging radiation delivery technique, such as swallowing sparing intensity modulation radiation therapy (IMRT) and proton radiotherapy.
* To compare the outcome of new radiation delivery techniques that are clinically introduced with the current standard in terms of radiation-induced toxicity, patient-rated symptoms and quality of life and in terms of locoregional tumour control and overall survival

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for curatively intended primary or postoperative radiotherapy will be included. At the first visit, patients are informed about the standard follow up program by the treating physician.

Exclusion Criteria:

* All patients planned for palliative radiotherapy will not be included in the SFP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with head and neck cancer planned for curatively intended primary or postoperative radiotherapy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2007-03; Primary Completion 2025-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Late toxicity | At 6 months after last day of completion of treatment
  Late toxicity

SECONDARY OUTCOMES:
Change in acute toxicity | At 1,2,3,4,5,6,7 (= during radiation therapy) and 12 weeks (= 6 weeks after completion of treatment) after first day of radiation therapy
  Change in acute toxicity
Change in patient-rated quality of life | At 6,12,18,24,36,48,60 months after completion of treatment
  Change in patient-rated quality of life
Overall survival | At 1,2,3,4 and 5 years after completion of treatment
  Overall survival
Change in locoregional tumour control | At 1,2,3,4 and 5 years after completion of treatment
  Change in locoregional tumour control
Laryngo-oesophageal dysfunction-free survival | At 1,2,3,4 and 5 years after completion of treatment
  Laryngo-oesophageal dysfunction-free survival
Change in patient-rated symptoms | At 1,2,3,4,5,6,7 (= during radiation therapy) and 12 weeks (= 6 weeks after completion of treatment) after first day of radiation therapy
  Change in patient-rated symptoms
Late toxicity | At 12 months after last day of completion of treatment
  Late toxicity
Late toxicity | At 18 months after last day of completion of treatment
  Late toxicity
Late toxicity | At 24 months after last day of completion of treatment
  Late toxicity
Late toxicity | At 36 months after last day of completion of treatment
  Late toxicity
Late toxicity | At 48 months after last day of completion of treatment
  Late toxicity
Late toxicity | At 60 months after last day of completion of treatment
  Late toxicity
Thyroid Stimulating Hormone (TSH) | At baseline and at 6, 12, 18, 24, 36, 48 and 60 months after completion of radiation therapy.
  TSH levels (mU/L) measured in blood
Free Thyroxine-4 (FT4) | At baseline and at 6, 12, 18, 24, 36, 48 and 60 months after completion of radiation therapy.
  FT4 levels (pmol/L) measured in blood

CONTACTS AND LOCATIONS:
Overall Officials: J.A. Langendijk, Prof. Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No